CLINICAL TRIAL: NCT00404898
Title: NYU/Bellevue Red Cross WTC Health Impacts Research Registry
Brief Title: NYU/Bellevue WTC Health Impacts Research Registry
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 06-01; NCT01751711 (obsolete NCT alias)
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Exposure to World Trade Center Dust
Keywords: World Trade Center dust

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The American Red Cross has funded a multidisciplinary, comprehensive evaluation and treatment program for target individuals with suspected World Trade Center (WTC)-related health problems. The populations served consist predominantly of a) local residents who were impacted by the disperion of the WTC dusts and fumes, b) individuals involved in cleaning and debris removal of local commercial spaces, and c) responders to the WTC collapse. These populations are recruited from past and ongoing programs that we have developed as well as from ongoing collaborations with community organizations that include: the Beyond Ground Zero Network, 9/11 Environmental Action committee, and the WTC Residents Coalition. In addition, there is collaboration with the Charles B. Wang Community Health Center and the centers involved in the ongoing WTC Workers and Volunteer Medical Screening and Monitoring Program. We would now like to access the data from this treatment program to create a NYU/Bellevue WTC Health Impacts Research Registry to increase knowledge about the health effects of exposure to World Trade Center dust.

ELIGIBILITY:
Target populations who will participate in the Bellevue Hospital Red Cross WTC Health Impacts Program will include:

* residents (children and adults) of Lower Manhattan communities at the time of the attacks, who remained or returned to their homes soon after the attacks
* individuals involved in debris removal in surrounding commercial and residential buildings,
* individuals involved in rescue, recovery and debris removal who have been previously screened through the World Trade Center Worker and Volunteer Medical Screening Program and are in need of continued treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The populations to be served will consist predominantly of a) local residents who were impacted by the dispersion of the WTC dusts and fumes, b) individuals involved in cleaning and debris removal of local commercial spaces, and c) responders to the WTC collapse. These populations will be recruited from past and ongoing programs that we have developed as well as from ongoing collaborations with community organizations that include: the Beyond Ground Zero Network, 9/11 Environmental Action committee, and the WTC Residents Coalition.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2007-12; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory Status | June 2020

SECONDARY OUTCOMES:
Mental Health Status | June 2020
General Health Status | June 2020

CONTACTS AND LOCATIONS:
Overall Officials: Joan Reibman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU School of Medicine/Bellevue Hospital, New York, New York, United States

REFERENCES:
- [Derived] Caplan-Shaw C, Kazeros A, Pradhan D, Berger K, Goldring R, Zhao S, Liu M, Shao Y, Fernandez-Beros ME, Marmor M, Levy-Carrick N, Rosen R, Ferri L, Reibman J. Improvement in severe lower respiratory symptoms and small airway function in World Trade Center dust exposed community members. Am J Ind Med. 2016 Sep;59(9):777-87. doi: 10.1002/ajim.22642. PMID 27582480